CLINICAL TRIAL: NCT07145112
Title: A Phase 1 Safety and Feasibility Study of Laser Interstitial Thermal Therapy (LITT) Followed by Lomustine (CCNU) for Recurrent Glioblastoma in Adults
Brief Title: Laser Interstitial Thermal Therapy (LITT) and Lomustine (CCNU) for Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC321; P30CA093373 (NIH); NCI-2025-06916 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2352196 (Other: UC Davis IRB)
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Laser interstitial thermal therapy (LITT) + Lomustine (CCNU) (Experimental): Laser interstitial thermal therapy (LITT) + Lomustine (CCNU)
  Interventions: Procedure: Laser interstitial thermal therapy; Drug: Lomustine

INTERVENTIONS:
Procedure: Laser interstitial thermal therapy — MRI guided laser
  Other Names: LITT
Drug: Lomustine — Given orally (PO)
  Other Names: CCNU, Gleostine

SUMMARY:
This is a phase 1 study evaluating the safety and feasibility of laser interstitial thermal therapy (LITT) followed by lomustine (CCNU) for recurrent glioblastoma in adults. The primary aim is to evaluate the safety of the combination of LITT plus lomustine based on the assessment of treatment-related adverse events and the feasibility of completing LITT + lomustine in the proposed timeframe. The secondary aim is to assess overall survival for up to 2 years after the first dose of lomustine.

DETAILED DESCRIPTION:
The LITT procedure is performed per standard of care under general anesthesia using a stereotactic neurosurgical approach where a laser catheter is precisely inserted into the tumor under MRI guidance. Real-time MRI thermometry is used to ensure controlled tumor ablation while minimizing damage to adjacent structures. Patients typically undergo postoperative MRI to assess treatment response, and most can be discharged within 24-48 hours, facilitating early initiation of adjuvant therapy.

Approximately 7 days following LITT, lomustine is administered per standard of care on Day 1 for a total of one cycle.

Participants will be monitored for serious and non-serious adverse events (AE) starting from initiation of LITT per institutional practices. All follow-up is based on standard of care for LITT and lomustine.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed World Health Organization (WHO) 2021 defined glioblastoma. A pathology report constitutes adequate documentation of histology for study inclusion.
2. Radiographic demonstration of disease progression following prior therapy.
3. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as the patient has recovered from surgery. Evaluable or measurable disease following resection of recurrent tumor is not mandated for eligibility into the study.
4. Prior standard radiation for glioblastoma (short course 40 Gy, standard 60 Gy, and proton therapy are allowed).
5. Patients must have recovered from the effects of prior therapy.
6. The following listed agents/interventions must have been discontinued for their respective time period prior to enrollment:

   1. Four weeks from cytotoxic agents (3 weeks from procarbazine, 3 weeks from vincristine, and 4 weeks from temozolomide);
   2. Four weeks or 5 drug half-lives (whichever is shorter) from any investigational agent; two weeks or 5 drug half-lives (whichever is shorter) from non-cytotoxic agents (e.g. Accutane, thalidomide);
   3. Twelve weeks from radiotherapy to minimize the potential for MRI changes related to radiation necrosis that might be misdiagnosed as progressive disease, or 4 weeks if a new lesion, relative to the pre-radiation MRI, develops that is outside the primary radiation field;
7. Patients must have the following laboratory parameters ≤ 14 days prior to registration:

   a. adequate bone marrow function defined by: i. white blood cells (WBC) ≥ 3 × 109/L , ii. absolute neutrophil count (ANC) ≥ 1.5 × 109/L , iii. platelet count of ≥ 100 × 109/L , and iv. hemoglobin ≥ 9 gm/dL b. adequate liver function defined by i. alanine transaminase (ALT, SGPT) and aspartate transaminase (AST/SGOT) < 3× institutional upper limit of normal (ULN), ii. alkaline phosphatase < 2× ULN, and iii. bilirubin < 1.5 mg/dL c. adequate renal function defined by calculated creatinine clearance ≥ 60 mL/min (see Appendix)
8. Karnofsky performance status (KPS) ≥ 50 (see Appendix).
9. Individuals of childbearing potential or those with partners of childbearing potential must agree to use adequate methods of contraception for the duration of study participation (including dosing interruptions) and for up to 3.5 months after the last study treatment; or be surgically sterilized.
10. Patients on the following medications are allowed:

    1. Anticoagulants: Patients on stable dose anticoagulants (e.g. warfarin in-range international normalized ratio [INR], low molecular-weight heparin)
    2. Patients are allowed to take aspirin, clopidogrel, ticlopidine, Aggrenox, ibuprofen and other NSAIDS.
11. Patients must be willing to forego other cytotoxic and non-cytotoxic drug therapy for glioblastoma while enrolled in the study.
12. Able to swallow oral medication.
13. Patients ≥18 years of age at time of consent.
14. Ability to understand and willingness to sign an informed consent form (ICF).
15. Ability and stated willingness to adhere to the study visit schedule and protocol procedures/requirements, including periodic blood sampling and study related assessments

Exclusion Criteria:

1. Patients who are not surgical candidates for stereotactic biopsy or laser ablation.
2. Prior treatment with nitrosourea agents (e.g. lomustine [CCNU], carmustine [BCNU], nimustine [ACNU]).
3. Prior treatment with polifeprosan 20 with carmustine wafer.
4. Prior treatment with bevacizumab.
5. Patients who have received any investigational agents ≤ 4 weeks or 5 drug half-lives (whichever is shorter) prior to commencing study treatment.
6. Evidence of recent hemorrhage on baseline MRI of the brain with the following exceptions: (1) presence of hemosiderin, (2) resolving hemorrhagic changes related to surgery, or (3) presence of punctate hemorrhage in the tumor.
7. History of intracerebral abscess within 6 months prior to Day 1.
8. Major surgical procedure, open biopsy, or significant traumatic injury ≤ 28 days prior to Day 1, or anticipation of the need for a major surgical procedure during the course of the study.
9. Serious non-healing wound, ulcer, or bone fracture.
10. Pregnancy (positive pregnancy test) or lactation.
11. Known hypersensitivity to any component of lomustine (CCNU).
12. Uncontrolled intercurrent illness or unstable systemic disease, including, but not limited to, ongoing or active infection, uncontrolled hypertension, or serious cardiac arrhythmia requiring medication that would interfere with participant safety or limit compliance with the study requirements.
13. Unable to undergo an MRI with contrast.
14. Known allergy to nitrosoureas (e.g., lomustine, carmustine, nimustine).
15. Any condition that in the opinion of the investigator would interfere with the participant's safety or compliance while on trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety of the combination of Laser Interstitial Thermal Therapy (LITT) and lomustine in patients with recurrent glioblastoma. | Up to 6 weeks after first dose of lomustine
  Number of treatment related adverse events, grade 3 and 4 using Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Tolerability of the combination of Laser Interstitial Thermal Therapy (LITT) and lomustine in patients with recurrent glioblastoma. | Up to 7 days post laser uinterstitial thermal therapy
  Percentage of participants completing LITT and receiving 1 dose of lomustine within the proposed timeframe (e.g., 7 days).

SECONDARY OUTCOMES:
Overall survival | Up to 2 years following first dose of lomustine.
  Median time of presentation to date of death or censored at last follow-up date.

CONTACTS AND LOCATIONS:
Overall Officials: Orwa Aboud, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States